CLINICAL TRIAL: NCT00275379
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Exploratory Study of Orally Administered ERB-041 in Subjects With Active Interstitial Cystitis
Brief Title: Study Evaluating Orally Administered ERB-041 in Subjects With Active Interstitial Cystitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A4-109; B2381036 (Other: Pfizer)
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Cystitis, Interstitial
Keywords: Cystitis
MeSH Terms: conditions — Cystitis, Interstitial; Cystitis | interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-design, exploratory study of orally administered ERB-041 in subjects with active IC. The primary objectives of this study will be to investigate ERB-041's activity on levels of urinary APF, explore the gene expression response in peripheral blood mononuclear cells (PBMC), and to evaluate the safety of ERB-041 in women with active IC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects seeking medical treatment for symptoms consistent with IC that have been ongoing for > 9 months or seeking medical treatment for a previous documented diagnosis of IC
* Subjects who are not surgically sterile or postmenopausal (amenorrheic > 12 months) must agree and commit to the use of a medically acceptable, highly-effective (i.e. double-barrier or IUD), non-hormonal form of birth control during the study and for 30 days after the last dose of test

Exclusion Criteria:

* Use of herbal supplements (except for a daily multivitamin/mineral supplement not containing herbal components)
* History of cancer (other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer) with less than 5 years documentation of a disease-free state
* Vaginitis or vaginal infection within 1 month before randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Safety
Levels of urinary antiproliferative factor (APF)
Peripheral blood mononuclear cell (PBMC) gene expression profiles

SECONDARY OUTCOMES:
Serum and urinary biomarkers of IC
Clinical Activity:
Global Response Assessment (GRA)
O'Leary-Sant IC Symptom (ICSI) and Problem (ICPI) Index
Pelvic Pain and Urinary/Frequency (PUF) Symptom Scale
Female Sexual Function Index (FSFI)
Voiding Diary

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Monitor, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com
Locations (14):
- United States (11):
  - Glendora, California
  - Redding, California
  - San Diego, California
  - Aventura, Florida
  - Kansas City, Kansas
  - Jackson, Michigan
  - Springfield, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Temple, Texas
  - Mountlake Terrace, Washington
- Baden, Austria
- Germany (2):
  - Homburg/Saar
  - Münster